CLINICAL TRIAL: NCT01958255
Title: Community Based Tobacco Cessation Programme
Brief Title: Community Based Tobacco Cessation Programme Mumbai
Acronym: CBTCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Associate Professor and Physician, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TMHPO912
Record Dates: First submitted 2013-09-27; First posted 2013-10-09 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Tobacco Smoking Behavior
Keywords: tobacco quit rates
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tobacco cessation counseling (Other): planned intervention for tobacco cessation counseling
  Interventions: Behavioral: planned intervention for tobacco cessation counseling

INTERVENTIONS:
Behavioral: planned intervention for tobacco cessation counseling — game session for rapport building followed by group discussion and tobacco cessation counseling

SUMMARY:
The aim of this project was to provide tobacco cessation services to the women at the community level at their door steps and thus establish a model community based tobacco cessation programme which could be replicated in other communities and could be taken up by National Tobacco Control Programme (NTCP), in future.

DETAILED DESCRIPTION:
The study was extended over a period of one year. There were 3 interventions given at the interval of 3 months each. The post intervention questionnaire regarding knowledge, attitude and practices was planned filled at the end of the programme i.e. 9th to 12th month from start of the programme. A community based tobacco cessation programme, which has the potential of being first of its kind, for women, was planned by the department of Preventive Oncology for the women in a geographical community in and around Mankhurd in Mumbai,for providing tobacco cessation counseling services. Doorstep services were provided to these women as they were unlikely to avail the tobacco cessation services at the clinic in TMH since their priority is managing household chores and caretaking of their family. The selected community was a part of women cancer screening programme namely; Tata Memorial Hospital Mobile Outreach Programme (TMH-MOP). The women who were current tobacco users at the time of screening under TMH-MOP were enrolled for this study.The women were intervened thrice at an interval of 3 months each and tobacco cessation counseling was provided at each intervention. The post intervention data was collected at the end of all the 3 counseling sessions. Sessions were held for rapport building with the participant women. Questionnaire were filled to record the information on the details of different forms of tobacco usage, factors responsible for initiation and continuation of tobacco use, pre-intervention and post-intervention knowledge, attitudes and practices regarding tobacco habits and severity of tobacco use (Fagerstroms scale). This programme was aimed at creating awareness and educating women regarding the health hazards of tobacco use, at the community level, at their door step.

ELIGIBILITY:
Inclusion Criteria:

all current tobacco users at the time of screening under TMH-MOP project

Exclusion Criteria:

All those who refused to participate and those who could not be contacted during the study period

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To assess tobacco quit rates | Baseline and 12 months
  The participant women were intervened thrice for counseling about quitting tobacco and quit rates were assessed at the end of one year

SECONDARY OUTCOMES:
To assess pre-intervention knowledge, attitude and practices about tobacco use. | baseline
  A questionnaire to assess the baseline knowledge, attitude and practices about tobacco use by participant women was filled during first intervention
To assess post-intervention knowledge, attitude and practices of tobacco use by participant women. | 9 month and 12 month
  A questionnaire to assess the baseline knowledge, attitude and practices about tobacco use by participant women was filled during post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A Mishra, M.D.PSM, Principal Investigator — Tata Memorial Hospital, Parel, Mumbai,India
Locations (1):
- Tata Memorial Hospital, Parel, Mumbai, Maharashtra, India